CLINICAL TRIAL: NCT05825339
Title: Absolute Flow for Ischemia With No Obstructive Coronary Arteries
Acronym: AF-INOCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Fernando Alfonso, Principal Investigator, Spanish Society of Cardiology
Other Study IDs: ES01100023
Record Dates: First submitted 2023-03-28; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Coronary Microvascular Dysfunction; Coronary Microvascular Disease; Angina, Stable
Keywords: Microvascular dysfunction; Coronary circulation; Myocardial ischemia Diagnosis; Coronary flow
MeSH Terms: conditions — Microvascular Angina; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary Flow Reserve — Diagnostic of Microvascular Coronary Dysfunction using continuous thermodilution flow reserve
  Other Names: Absolute Flow

SUMMARY:
The main objective is to prospectively validate the capacity of continuous thermodilution coronary flow reserve (CFRflow) as a predictor of the presence of angina measured by SAQ7 in patients with INOCA at 3 months. Secondary objectives include identifying hemodynamic factors related to the persistence of angina at 3 and 12 months, identifying clinical factors associated with the persistence of angina, establishing the prevalence of patients with coronary microvascular dysfunction within the cohort of INOCA patients, identifying predictors of major cardiovascular events at 12 months, validating the pathological value of MMR and establishing the pathological value of AF measured in ml/min. The study also aims to evaluate the concordance between measures of the coronary microvascular function obtained by continuous thermodilution and bolus thermodilution, as well as their concordance with clinical characteristics.

DETAILED DESCRIPTION:
Invasive study of microvascular function has become highly relevant for the diagnosis of alterations in coronary physiology for diagnostic, prognostic, and therapeutic purposes. Currently, the microvascular resistance index (IMR) is considered the gold standard for invasive diagnosis of coronary microvascular function, with a recommendation of 2A in the current clinical practice guidelines of the European Society of Cardiology. In recent years, technical innovation has allowed for the measurement of absolute coronary flow (AF) and minimal microvascular resistance (MMR) using continuous thermodilution, enabling the determination of quantitative flow and resistance units. However, the main limitation is the absence of reference values.

Objectives:

The main objective is to prospectively validate the capacity of CFRflow as a predictor of the presence of angina measured by SAQ7 in patients with INOCA at 3 months. Secondary objectives include identifying hemodynamic factors related to the persistence of angina at 3 and 12 months, identifying clinical factors related to the persistence of angina, establishing the prevalence of patients with coronary microvascular dysfunction within the cohort of INOCA patients, identifying predictors of major cardiovascular events at 12 months, validating the pathological value of MMR and establishing the pathological value of AF measured in ml/min. The study also aims to evaluate the concordance between measures of the coronary microvascular function obtained by continuous thermodilution and bolus thermodilution, as well as their concordance with clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, and
* Clinical indication for coronary angiography and in whom the use of microvascular function diagnosis by pressure guide is considered clinically necessary.
* Clinical diagnosis of typical or atypical angina.
* Coronary arteries without lesions or with epicardial lesions <50% by visual estimation or fractional flow reserve (FFR)>0.80.
* Absence of clinical or anatomical contraindications for the study of microvascular function.

Consent for participation in the study prior to information and consent form signature.

Exclusion Criteria:

* Decompensated heart failure or cardiogenic shock.
* Admission due to Acute Coronary Syndrome with an elevation of markers in the month prior to inclusion.
* Indication for coronary angioplasty.
* Severe pulmonary hypertension.
* Obstructive hypertrophic cardiomyopathy.
* Severe valvular disease.
* Previous allergy or intolerance to adenosine or adenosine triphosphate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a clinical indication for diagnostic study of coronary microvascular function due to angina without obstructive coronary lesions.
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Angina Status | At inclusion
  Angina Status assessed by Seattle Angina Questionnaire (SAQ).The total score is also transformed into a scale from 0 to 100, where a higher score indicates better angina-related quality of life.

SECONDARY OUTCOMES:
Quality of life at 3 months | 3 months
  Quality of life status in patients at 3 months post-diagnosis measured by the Seattle Angina Questionnaire (SAQ).The total score is also transformed into a scale from 0 to 100, where a higher score indicates better angina-related quality of life.
Accuracy of continuous thermodilution coronary flow reserve (CFR) measured by Youden Index = Sensitivity + Specificity - 1 | At inclusion
  Continuous thermodilution measured CFR flow and minimal microvascular resistance (MMR flow).

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rivero F, Gutierrez-Barrios A, Gomez-Lara J, Fuentes-Ferrer M, Cuesta J, Keulards DCJ, Pardo-Sanz A, Bastante T, Izaga-Torralba E, Gomez-Hospital JA, Garcia-Guimaraes M, Pijls NHJ, Alfonso F. Coronary microvascular dysfunction assessed by continuous intracoronary thermodilution: A comparative study with index of microvascular resistance. Int J Cardiol. 2021 Jun 15;333:1-7. doi: 10.1016/j.ijcard.2021.03.005. Epub 2021 Mar 5. PMID 33684380
- [Result] de Vos A, Jansen TPJ, van 't Veer M, Dimitriu-Leen A, Konst RE, Elias-Smale S, Paradies V, Rodwell L, van den Oord S, Smits P, van Royen N, Pijls N, Damman P. Microvascular Resistance Reserve to Assess Microvascular Dysfunction in ANOCA Patients. JACC Cardiovasc Interv. 2023 Feb 27;16(4):470-481. doi: 10.1016/j.jcin.2022.12.012. PMID 36858668
- [Result] Gallinoro E, Bertolone DT, Fernandez-Peregrina E, Paolisso P, Bermpeis K, Esposito G, Gomez-Lopez A, Candreva A, Mileva N, Belmonte M, Mizukami T, Fournier S, Vanderheyden M, Wyffels E, Bartunek J, Sonck J, Barbato E, Collet C, De Bruyne B. Reproducibility of bolus versus continuous thermodilution for assessment of coronary microvascular function in patients with ANOCA. EuroIntervention. 2023 Jun 5;19(2):e155-e166. doi: 10.4244/EIJ-D-22-00772. PMID 36809253
- [Result] De Bruyne B, Pijls NHJ, Gallinoro E, Candreva A, Fournier S, Keulards DCJ, Sonck J, Van't Veer M, Barbato E, Bartunek J, Vanderheyden M, Wyffels E, De Vos A, El Farissi M, Tonino PAL, Muller O, Collet C, Fearon WF. Microvascular Resistance Reserve for Assessment of Coronary Microvascular Function: JACC Technology Corner. J Am Coll Cardiol. 2021 Oct 12;78(15):1541-1549. doi: 10.1016/j.jacc.2021.08.017. PMID 34620412
- [Result] Jansen TPJ, Konst RE, Elias-Smale SE, van den Oord SC, Ong P, de Vos AMJ, van de Hoef TP, Paradies V, Smits PC, van Royen N, Damman P. Assessing Microvascular Dysfunction in Angina With Unobstructed Coronary Arteries: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Oct 5;78(14):1471-1479. doi: 10.1016/j.jacc.2021.08.028. PMID 34593129